CLINICAL TRIAL: NCT05720221
Title: Adalimumab Versus Ustekinumab in Management of Inflammatory Bowel Disease in Egyptian Patients
Brief Title: Biologics in Management of Inflammatory Bowel Disease in Egyptian Patients
Status: Completed | Type: Observational
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Eman Magdy El-sayed El-yamany, Teaching assistant at pharmacy practice department, Faculty of Pharmacy, Helwan University
Other Study IDs: Biologics in IBD
Record Dates: First submitted 2022-12-02; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: IBD
Keywords: Ustekinumab; Adalimumab; IBD; Stelara; Humira

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adalimumab group: Patients receive adalimumab (Humira) at an induction dose of 160/80 mg (week 0 and 2) and at a maintenance dose of 40 mg every other week.
  The efficacy of the drug will be assessed.
- Ustekinumab group: Patients receive ustekinumab (Stelara) through intravenous infusion with a weight based dose for treatment induction, followed by a subcutaneous dose injection with a fixed dose (90 mg) for maintenance every 8 weeks.
  The efficacy of the drug will be assessed.

SUMMARY:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), is a chronic inflammatory relapsing disorder affecting the gastrointestinal tract and is characterized by a progressive and unpredictable disease course.The two goals of therapy are the achievement of remission (induction) and the prevention of disease flares (maintenance). Medical therapy for IBD has advanced dramatically in the last decade with the introduction of targeted biologic therapies including infliximab,adalimumab and ustekinumab.There is paucity of head-to-head studies comparing the effectiveness of ustekinumab and adalimumab in inflammatory bowel disease patients especially in Egyptian population which prompted this study to be conducted.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), is a chronic inflammatory relapsing disorder affecting the gastrointestinal tract and is characterized by a progressive and unpredictable disease course. There has been a global rise in the incidence of IBD over the last few decades, in 2017; there were 6.8 million cases of IBD globally. The age-standardized prevalence rate increased from 79.5 per 100, 000 population in 1990 to 84.3 per 100, 000 population in 2017. The annual incidence of Crohn's disease is 5.0 per 100,000 person-years in Asia and the Middle East, whereas incidence rates of ulcerative colitis are 6.3 per 100,000 person-years in Asia and the Middle East. The male-to-female ratio is approximately 1:1 for ulcerative colitis and Crohn's disease, with females having a slightly greater incidence. Both diseases are most commonly diagnosed in young adults (i.e., late adolescence to the third decade of life). Although the etiology of IBD remains largely unknown, it involves a complex interaction between the genetic, environmental or microbial factors and the immune responses. The symptoms of IBD include: diarrhea (often loose and watery with Crohn's disease or bloody with ulcerative colitis), severe or chronic cramping pain in the abdomen, loss of appetite leading to weight loss, fatigue, fever, rectal bleeding, joint pain and skin problems, such as rashes. The two goals of therapy are the achievement of remission (induction) and the prevention of disease flares (maintenance). Medical therapy for IBD has advanced dramatically in the last decade with the introduction of targeted biologic therapies including infliximab,adalimumab and ustekinumab, the optimization of older therapies, including rugs such as immunomodulators and 5-aminosalicylic acid (5-ASA), and a better understanding of the mucosal immune system and the genetics involved in the pathogenesis of IBD.

Adalimumab (ADA) is a monoclonal immunoglobulin G1 antibody that binds with high affinity and specificity to human TNF. ADA is an anti-TNF agent that has been shown to be effective in inducing and maintaining remission in patients with IBD at an induction dose of 160/80 mg (week 0 and 2) and at a maintenance dose of 40 mg every other week. The efficacy of adalimumab as a second-line therapy has also been documented for patients with loss of response or intolerance to infliximab. Ustekinumab, the monoclonal antibody to the p40 subunit of interleukin IL-12 and IL-23, has been approved in 2016 for the use in patients with moderate to severe active Crohn's disease (CD) and it was approved by the US Food and Drug Administration (FDA) for the treatment of moderate to severe ulcerative colitis in October 2019. The administration of ustekinumab for induction is intravenous and weight-based followed by a subcutaneous dose injection with a fixed dose (90 mg) for maintenance.

There is paucity of head-to-head studies comparing the effectiveness of ustekinumab and adalimumab in inflammatory bowel disease patients especially in Egyptian population which prompted this study to be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Age:18 year old or more.
* Gender: both male and female patients.
* Patients with IBD diagnosis established by clinical, laboratory and endoscopic findings.
* Moderate to severe inflammatory bowel disease patients.

Exclusion Criteria:

* Age less than 18 years.
* Malignancy.
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A comparative, prospective, observational cohort study will be conducted. Patients will be selected according to the inclusion and the exclusion criteria.
  Patient's clinical data will include: age, sex, surgical history and associated comorbidities.
  The patients will be divided into two groups:
  Group 1 is adalimumab group Group 2 is ustekinumab group The follow up duration will be six months for each patient. Follow up duration: six months.
  Parameters will be monitored in both groups during the study period as:
  C-reactive protein (CRP) , complete blood count (CBC) and clinical scores.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving the clinical response after 4 months from baseline | Baseline to four months.
  Percentage of patients achieving the clinical response will be assessed, the clinical response defined as reduction of at least 3 points of Harvey Bradshaw Index (HBI) from baseline (in chrons disease) and reduction of at least 2 points of Partial Mayo Score (PMS) from baseline (in ulcerative colitis). [time frame baseline to 4 months]

SECONDARY OUTCOMES:
Percentage of patients achieving the clinical remission after 4 months from baseline | Baseline to six months.
  Percentage of patients achieving the clinical remission that defined as Harvey Bradshaw Index (HBI) < 5 points (in chrons disease patients) and Partial mayo score (PMS) < 2 points (in ulcerative colitis patients).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of pharmacy-Helwan University, Cairo, Egypt

REFERENCES:
- [Background] Baumgart DC, Carding SR. Inflammatory bowel disease: cause and immunobiology. Lancet. 2007 May 12;369(9573):1627-40. doi: 10.1016/S0140-6736(07)60750-8. PMID 17499605
- [Background] GBD 2017 Inflammatory Bowel Disease Collaborators. The global, regional, and national burden of inflammatory bowel disease in 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Gastroenterol Hepatol. 2020 Jan;5(1):17-30. doi: 10.1016/S2468-1253(19)30333-4. Epub 2019 Oct 21. PMID 31648971
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Langholz E. Current trends in inflammatory bowel disease: the natural history. Therap Adv Gastroenterol. 2010 Mar;3(2):77-86. doi: 10.1177/1756283X10361304. PMID 21180592
- [Background] Zhang YZ, Li YY. Inflammatory bowel disease: pathogenesis. World J Gastroenterol. 2014 Jan 7;20(1):91-9. doi: 10.3748/wjg.v20.i1.91. PMID 24415861
- [Background] Amezaga AJ, Van Assche G. Practical Approaches to "Top-Down" Therapies for Crohn's Disease. Curr Gastroenterol Rep. 2016 Jul;18(7):35. doi: 10.1007/s11894-016-0507-z. PMID 27184044
- [Background] Pithadia AB, Jain S. Treatment of inflammatory bowel disease (IBD). Pharmacol Rep. 2011;63(3):629-42. doi: 10.1016/s1734-1140(11)70575-8. PMID 21857074
- [Background] Hinojosa J, Munoz F, Martinez-Romero GJ. Relationship between Serum Adalimumab Levels and Clinical Outcome in the Treatment of Inflammatory Bowel Disease. Dig Dis. 2019;37(6):444-450. doi: 10.1159/000499870. Epub 2019 Apr 30. PMID 31039560
- [Background] Guidi L, Pugliese D, Armuzzi A. Update on the management of inflammatory bowel disease: specific role of adalimumab. Clin Exp Gastroenterol. 2011;4:163-72. doi: 10.2147/CEG.S14558. Epub 2011 Jul 15. PMID 21904462
- [Background] Restellini S, Afif W. Update on TDM (Therapeutic Drug Monitoring) with Ustekinumab, Vedolizumab and Tofacitinib in Inflammatory Bowel Disease. J Clin Med. 2021 Mar 17;10(6):1242. doi: 10.3390/jcm10061242. PMID 33802816
- [Background] Ahmed Z, Venkata K, Zhang N, Malik TA. Comparative Effectiveness of Ustekinumab Versus Adalimumab in Induction of Clinical Response and Remission in Crohn's Disease: Experience of a Real-World Cohort at a Tertiary Care Inflammatory Bowel Disease Referral Center. Gastroenterology Res. 2019 Oct;12(5):245-251. doi: 10.14740/gr1194. Epub 2019 Oct 4. PMID 31636774
- [Background] Ochsenkuhn T, Tillack C, Szokodi D, Janelidze S, Schnitzler F. Clinical outcomes with ustekinumab as rescue treatment in therapy-refractory or therapy-intolerant ulcerative colitis. United European Gastroenterol J. 2020 Feb;8(1):91-98. doi: 10.1177/2050640619895361. Epub 2019 Dec 12. PMID 32213052